CLINICAL TRIAL: NCT00423566
Title: A Phase I Study of the Safety and Immunogenicity of a Recombinant MVA Vaccine Encoding a Secreted Antigen From M. Tuberculosis, Antigen 85A, Delivered Intradermally by a Needle Injection in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB002
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2006-12

CONDITIONS: Tuberculosis
Keywords: Mycobacterium tuberculosis; 85A antigen; Recombinant Modified Vaccinia virus Ankara; Phase I study; Immunogenicity
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A; Tuberculosis Vaccines

INTERVENTIONS:
Biological: MVA85A (Tuberculosis vaccine)

SUMMARY:
This study is to assesss the safety and immunogenicity of vaccine based on Modified Vaccinia Ankara (MVA) expressing the 85A antigen (from Mycobacterium. tuberculosis). This vaccine is delivered intrdermally by a needle injection in healthy volunteers.

DETAILED DESCRIPTION:
1. This is a phase I study to assesss the safety and immunogenicity a recombinant MVA encoding a secreted antigen from Mycobacterium. tuberculosis Antigen 85A, delivered intrdermally by a needle injection in healthy BCG naive volunteers.
2. Selection of volunteers

   Volunteers for the study will be recruited through advertisements. Each volunteer will have received an information sheet concerning the study and will have agreed to participate in writing. Volunteers will be given at least 48 hours between reading the information leaflet and agreeing to participate. Female volunteers will be told of the theoretical risk of congenital anomaly should they become pregnant during the study and only those who undertake to take precautions to avoid pregnancy during the study period will be eligible. Volunteers will give signed consent for their GP's to be notified about their participation in the trial. The GP will be faxed a letter on the day of screening and asked to reply if they know of a reason why the volunteer should not take part. The signed consent form will also be faxed with the letter.
3. Screening

   Volunteers will be asked to sign the informed consent form for screening. The following will be performed:
   * Medical history and examination
   * Laboratory evaluations - including clinical chemistry, haematology, HLA typing, anti-vaccinia antibodies, anti-HBV antibodies, anti-HCV antibodies, anti-HIV antibodies
   * Heaf test - to exclude prior exposure to TB
   * Urinalysis and urine pregnancy test if female
4. Inclusion Criteria

   * Healthy adult aged 18-45 years.
   * Normal medical history and physical examination.
   * Normal urine dipstick, blood count, liver enzymes, and creatinine.
5. Exclusion Criteria

   1. Exposure to TB/BCG vaccination at any point. Previous residence in a TB endemic area.
   2. Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness, psychiatric disorder, drug or alcohol abuse.
   3. Oral or systemic steroid medication or the use of immunosuppressive agents.
   4. Positive HIV antibody test, HCV antibody test or positive HBV serology except post-vaccination.
   5. Positive Heaf test
   6. Confirmed pregnancy
   7. Previous MVA immunisations
6. Withdrawal Criteria

   1. Withdrawal of consent by subject for any reason
   2. Loss to follow-up
   3. Non-compliance with study procedures
   4. Protocol violation
   5. Serious adverse event (as defined in Appendix 3)
   6. Any other reason at discretion of the Principal Investigator
   7. Confirmed pregnancy during study period

      7 Immunisation

      On Day 0 and Day 21, subjects will receive a single intradermal injection of 5 x 107pfu in 0.1ml over the deltoid muscle. Subjects will be observed for an hour after all immunisations. Vital signs will be monitored at 30 and 60 minutes post-immunisation. Local reactions at the site of administration will be evaluated at 60 minutes.

      A photograph of the injection site may be taken at 48 hours (with written consent). The injection site will be reviewed 7 days after each immunization.

      Blood will be taken at the following time points: At the screening visit*, prior to the first vaccination, *1 week after the first vaccination, prior to the second vaccination, *1 week after the second vaccination, 4 weeks, 8 weeks, *12 weeks and 24 weeks after the second vaccination. Up to 55 mls will be taken at any one time with the total being no more than 500 mls over the study period. *Samples taken on these dates will be tested for full blood count and biochemical screen. Immunological assays will be performed at all time points to determine vaccine immunogenicity. A pregnancy test will be performed on screening and each vaccination day prior to vaccination for female volunteers. Peripheral blood mononuclear cells will be prepared for cellular immunological assays to be performed without or following cryopreservation. Other serological measures of immune response, i.e. antibody titres, will be assayed on frozen plasma samples.

      At the end of the six month follow-up period, volunteers will be offered BCG immunisation. If they accept, imunological monitering will continue for a further six months. 50mls of blood will be taken for cellular immunological assays 1 week, 2 weeks, 1 month, 2 months, 3 months and 6 months after BCG immunisation.

      All blood tests will be taken within 1-3 days of the due date as described in the schedule above.

      8 Endpoints

      The occurance and severity of local side-effects. The occurance and severity of systemic side-effects. The induction of T cell responses (as measured by an interferon-gamma Elispot assay).

      Proliferation assays and cytotoxic T cell assays will be performed on strong CD4+ and CD8+ responses respectively.

      This study has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-45 years.
* Normal medical history and physical examination.
* Normal urine dipstick, blood count, liver enzymes, and creatinine.

Exclusion Criteria:

* Exposure to TB/BCG vaccination at any point. Previous residence in a TB endemic area.
* Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness, psychiatric disorder, drug or alcohol abuse.
* Oral or systemic steroid medication or the use of immunosuppressive agents.
* Positive HIV antibody test, HCV antibody test or positive HBV serology except post-vaccination.
* Positive Heaf test
* Confirmed pregnancy
* Previous MVA immunisations

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14
Dates: Start 2002-09; Study Completion 2003-07

PRIMARY OUTCOMES:
Local and systemic reactions will be monitored 30 and 60 minutes after administration.
A photograph of the injection will be taken at 48 hours and this injection site will be reviewed 7 days after each immunisation.
Blood will be taken: 1 week after the first vaccination, 1 week after the second vaccination and then at 4, 8, 12 and 24 weeks. The blood is used for a full blood count and biochemical screen.
Immunological assays are performed at all time points to determine vaccine imunogenicity (T cell responses are measured using an interferon-gamma Elispot assay).

SECONDARY OUTCOMES:
Immunological assays are performed at all time points to determine vaccine imunogenicity (T cell responses are measured using an interferon-gamma Elispot assay).

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, MD and PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom